CLINICAL TRIAL: NCT05698212
Title: Proof-of-Concept, Obs Study to Evaluate Accuracy of MetriDx Lab Developed Test (LDT) to Accurately Identify Endometriosis-specific Biological Markers Using Micro-fluidic Analysis of Cells Enabling Clinicians to Diagnose Endometriosis
Brief Title: Proof of Concept Study to Eval MetriDx Lab-developed Test to Identify Endometriosis-specific Bio Markers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hera Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HER001
Record Dates: First submitted 2022-11-29; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-11

CONDITIONS: Endometriosis; Diagnosis
Keywords: endometriosis; MetriDx; connexins; biological markers; micro-fluidic analysis; uterine tissue biopsy
MeSH Terms: conditions — Endometriosis; Disease

STUDY DESIGN:
Intervention Model Description: Two cohorts defined by confirmed diagnosis of endometriosis and further grouping by staging of endometriosis A third cohort of control participants who have not been suspected or diagnosed with endometriosis
Who Masked: Outcomes Assessor
Masking Description: The lab associates conducting the diagnosis tests are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Active Comparator): Endometriosis diagnosed at stage 1 or 2
  Interventions: Diagnostic Test: MetriDx
- Cohort 2 (Active Comparator): Endometriosis diagnosed at stage 3 or 4
  Interventions: Diagnostic Test: MetriDx
- Cohort 3 (Other): Control--Not suspected of having and absence of endometriosis confirmed by diagnostic test.
  This group has uterine tissue biopsy and laparoscopy for non-endometriosis indication, i.e. tubal ligation
  Interventions: Diagnostic Test: MetriDx

INTERVENTIONS:
Diagnostic Test: MetriDx — Biopsied tissue will be analyze by proprietary LDT, MetriDx, and compared to laparoscopy diagnostic report on record

SUMMARY:
This study is testing a way to diagnose endometriosis using a uterine tissue biopsy (similar to a pap smear) as opposed to undergoing laparoscopy surgery. The tissue is sent to lab for cellular analysis with a proprietary AI (artificial intelligence) technology.

DETAILED DESCRIPTION:
This study involves 2 visits to the site and possibly as outpatient surgical center, and the participant will be involved in the for as little as 1 day to as much as 60 days, mainly depending on scheduling of laparoscopy. Eligible participants in the active group will have history of endometriosis and will be having a laparoscopy for diagnosis within the next few weeks. Eligible participants in the control group will have no history of endometriosis but will need or have recently had a laparoscopy surgical procedure for a reasons such as tubal ligation.

The participant will have an uterine biopsy (similar to a pap smear) in the physician's office before the laparoscopy. The biopsied tissue will be sent to a special lab for analysis and diagnosis of endometriosis by an innovative proprietary procedure that analyses the cells of the tissue collected in the biopsy.

The results of the biopsy will be compared to the laparoscopy for accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and provide informed consent.
* Natural born female of childbearing potential.
* Age between 18 and 50, inclusive.
* Not pregnant at Visit 0 (screening) or Visit 1 (day of procedure).
* Free of systemic or pelvic disorder that, in the opinion of the investigator, may interfere with the tissue collection procedure, analysis of the tissue or increase the risk to subject.
* Must not have received excision or ablation surgical procedure or treatment, such as gonadotropin-releasing hormone (GnRH), for endometriosis within the past 12 months.
* For Cohort 1 and 2:

  * Suspected of having endometriosis, or previously diagnosed with endometriosis, and currently recommended for laparoscopic surgery by physician.
  * Must have laparoscopic surgery within 60 days after screening Visit 0 and any time after the endometrial biopsy is obtained on Visit 1 (including the same day), or a laparoscopy on record within the 12 months prior to Visit 0 for diagnosis only.
  * Surgical report from prior laparoscopy must indicate that endometriosis was not treated with surgical ablation or excision.
  * Subjects will be assigned to Cohort 1 or 2 based on diagnosis and staging results from laparoscopy.
* Or for Cohort 3:

  * Not suspected of having endometriosis
  * no previous diagnosis or symptoms of endometriosis, who have had a laparoscopy for another reason, such as tubal ligation or other abdominal procedure, within the past 12 months prior to screening Visit 0,
  * or laparoscopy to be completed within 60 days after screening Visit 0 and any time after the endometrial biopsy is obtained on Visit 1 (including the same day).
  * Surgeon's report must have no supplemental observations of endometriosis lesions or diagnosis. Subjects will be assigned to Cohort 3.

Exclusion Criteria:

* Younger than 18 or 51 years or older.
* Surgical history of hysterectomy.
* Has received excision or ablation surgical procedure or treatment, such as gonadotropin-releasing hormone (GnRH), for endometriosis within the past 12 months.
* Cohort 3: Prior diagnosis of endometriosis, or surgical note from prior laparoscopy that indicates endometriosis lesions were observed.
* Has a BMI 40 or above.
* Is currently taking a blood thinner medication.
* Currently, pregnant, breast feeding, or has given birth in the last 6 months.
* Diagnosed with HIV, AIDS, hepatitis A, B, or C, or has active malignancy.
* Has a complicating condition that would pose a hazard to tissue handling.
* Undergoing fertility or hormone therapy treatments.
* History or evidence of uterine fibroids.
* History of reproductive cancer.
* Has a condition that, in the opinion of the investigator, would confound tissue collection or analysis.
* Has an active pelvic infection or other infections contra-indicated for laparoscopy.
* Has participated in any interventional clinical trial in the previous 90 days in which an investigational drug was administered.
* Has a history of alcohol or illegal drug/substance abuse, or suspected alcohol or illegal drug/substance abuse in the past two years.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Natural born female
Enrollment: 75 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-03-25 (Estimated); Study Completion 2023-04-10 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 1 week after laparoscopy
  Endometriosis diagnosis

SECONDARY OUTCOMES:
Secondary Outcome | 1 week after laparoscopy
  Accurate staging of endometriosis
Tertiary Outcome | 1 week after providing menstrual effluent sample
  observe and explore any relationship between subject's estrogen and progesterone levels and MetriDx results.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra M Hurtado, MD, Principal Investigator — University of Texas Physicians Women's Center; Charles R Kirkham, MD, Principal Investigator — Corpus Christi Women's Clinic; Jacqueline A Robinson, MD, Principal Investigator — Valley OB-GYN Clinic
Locations (3):
- United States (3):
  - Valley OB-GYN Clinic, PC, Saginaw, Michigan
  - Corpus Christi Women's Center, Corpus Christi, Texas
  - University of Texas Physician's Women's Center--Memorial City, Houston, Texas

IPD SHARING:
Plan to Share IPD: No